CLINICAL TRIAL: NCT03261934
Title: Risk Assessment and Syndrome Evolution Models Combining Traditional Chinese Medicine and Modern Medicine Indicators for Chronic Atrophic Gastritis Malignant Transformation: a Registry Study
Brief Title: Risk Assessment and Syndrome Evolution Models for Chronic Atrophic Gastritis Malignant Transformation
Status: Recruiting | Type: Observational
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: The University of Science and Technology of China (Other); China Academy of Chinese Medical Sciences (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Dr. Xia Ding, Professor, Beijing University of Chinese Medicine
Other Study IDs: 81630080-CAG-REG
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Risk Assessment of Chronic Atrophic Gastritis Malignant Transformation
Keywords: Chronic Atrophic Gastritis; Malignant Transformation; Risk Assessment; Syndrome Evolution; Traditional Chinese Medicine; Registry Study
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Paraffin section of gastric mucosa
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Chronic atrophic gastritis (CAG) is acknowledged as the precancerous stage of gastric cancer (GC). The present study aims to developed risk assessment and syndrome evolution models of CAG malignant transformation events combining TCM indicators with modern medicine indicators. The proposed study is a registry study based participant survey conducted in 4 hospitals in Beijing, China. After obtaining informed consent, a total of 2000 study patients diagnosed with CAG will be recruited. 10-year follow-ups are carried out on-site in hospitals and off-site by telephone to track malignant transformation events.

DETAILED DESCRIPTION:
Chronic atrophic gastritis (CAG) is acknowledged as the precancerous stage of gastric cancer (GC). Active treatment of CAG is vital in arresting malignant transformation. Traditional Chinese medicine (TCM) has been widely used in treating CAG and preventing GC. To date, no study has been conducted to assess the risk and syndrome evolution features of CAG malignant transformation by establishing models combining both TCM and modern medicine indicators.

The present study aims to developed risk assessment and syndrome evolution models of CAG malignant transformation events combining TCM indicators with modern medicine indicators. The proposed study is a registry study based participant survey conducted in 4 hospitals in Beijing, China. After obtaining informed consent, a total of 2000 study patients diagnosed with CAG will be recruited. 10-year follow-ups are carried out on-site in hospitals and off-site by telephone to track malignant transformation events. Comparative analysis of prevalence of malignant transformation events and presenting TCM or modern medicine features in different groups is conducted using frequency analysis and chi-squared tests, and expressed with composition ratios. Correlation analysis of malignant transformation events and TCM or modern medicine factors will be performed using logistic regression, and multivariate Cox proportional hazard model respectively. Exploratory factor analysis, correspondence analysis, association rule analysis, hierarchical clustering analysis, and complex system entropy clustering analysis will also be performed respectively for validating features of syndrome evolution in CAG malignant transformation process.

Previous reports on modern medicine indicators based risk assessment model for ischemic stroke endpoint events exist, but no studies have been undertaken combining TCM features. The risk assessment model combining both TCM and modern medicine indicators has the potential to facilitate early warning, early intervention and early control of CAG malignant transformation. The syndrome evolution model will help evaluate the core TCM pathogenesis of CAG malignant transformation so as to promote optimization of treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

(1) 18-75 years of age; (2) Meeting diagnostic criteria of CAG after upper gastrointestinal endoscopy; (3) Willing to cooperate with data, tissue sample, and blood sample collection during recruitment; (4) Willing to respond truthfully and timely to researcher queries after recruitment, able to cooperate with data, tissue sample and blood sample collection during follow-ups; (5) Willing to sign informed consent.

Exclusion Criteria:

(1) Meeting past history of previous stomach surgery; (2) Unable to participate in data, tissue sample or blood sample collection for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter registry study conducted in 4 hopitals in Beijing, China, leaded by Beijing University of Chinese Medicine. According to the inclusion and exclusion criteria, 2000 eligible participants will be identified by screening CAG patients after beginning the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
malignant transformation events of chronic atrophic gastritis | 10 years follow-up
  The primary outcome measures will be the malignant transformation events of chronic atrophic gastritis, including gastric mucosal atrophy, intestinal metaplasia, gastric intraepithelial dysplasia, and gastric carcinoma, according to the definition given by "Chronic Gastritis Diagnosis and Treatment Consensus of China (version 2012)", as promulgated by the Society of Gastroenterology, Chinese Medical Association.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Dongzhimen Hospital, Beijing, Beijing Municipality
  - Wangjing Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No